CLINICAL TRIAL: NCT02657889
Title: Phase 1/2 Clinical Study of Niraparib in Combination With Pembrolizumab (MK-3475) in Patients With Advanced or Metastatic Triple-Negative Breast Cancer and in Patients With Recurrent Ovarian Cancer
Brief Title: Niraparib in Combination With Pembrolizumab in Patients With Triple-negative Breast Cancer or Ovarian Cancer
Acronym: TOPACIO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213363; 3000-PN162-01-001 (Other: Tesaro)
Record Dates: First submitted 2016-01-08; First posted 2016-01-18 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Neoplasms; Triple Negative Breast Cancer; Ovarian Cancer; Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Stage IV Breast Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: PARP inhibitor; PD-1; Niraparib; Pembrolizumab; Keynote; TOPACIO
MeSH Terms: conditions — Neoplasms; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Fallopian Tube Neoplasms | interventions — niraparib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- niraparib plus pembrolizumab (Experimental): Phase 1: Dose-escalation: ascending doses of niraparib up to 300mg/day orally (PO) on Days 1-21 and pembrolizumab 200mg intravenously (IV) on Day 1 of each 21-day cycle
  Phase 2: niraparib (recommended Phase 2 dose) in combination with pembrolizumab 200mg IV on Day 1 of each 21-day cycle
  Interventions: Drug: niraparib; Biological: pembrolizumab

INTERVENTIONS:
Drug: niraparib
Biological: pembrolizumab

SUMMARY:
This Phase 1/2 study will evaluate the safety and efficacy of combination treatment with niraparib and pembrolizumab (MK-3475) in patients with advanced or metastatic triple-negative breast cancer or recurrent ovarian cancer. (KEYNOTE-162)

ELIGIBILITY:
Main Inclusion Criteria:

* Patient has histologically proven advanced (unresectable) or metastatic cancer as outlined below according to study phase and disease type:

  1. Phase 1 patients (breast or ovarian cancer)

     * Patients with advanced or metastatic breast cancer must have disease that is HER2-negative, estrogen receptor-negative, and progesterone receptor-negative (ie, TNBC). Patients with advanced or metastatic disease may have up to 4 lines of cytotoxic therapy. Neoadjuvant and adjuvant therapies are not counted towards lines of therapy.
     * Patients must have any epithelial (ie, serous, endometroid, mucinous, clear cell) ovarian, fallopian tube, or primary peritoneal cancer. Patients must have experienced a response lasting at least 6 months to first-line platinum-based therapy but currently considered to have platinum-resistant disease per investigator's assessment (e.g, patient is not eligible for further platinum containing treatment). Patients may have received up to 5 lines of cytotoxic therapy for advanced or metastatic cancer. Neoadjuvant and adjuvant therapies are not counted towards lines of therapy.
  2. Phase 2 patients (breast or ovarian cancer)

     * Patients with advanced or metastatic breast cancer must have TNBC. Patients with advanced or metastatic disease may have received up to 2 lines of cytotoxic therapy. Adjuvant and/or neoadjuvant therapies are not counted in the number of lines of therapy. TNBC patients who have previously received platinum chemotherapy in the metastatic setting are allowed to enroll in the study as long as they did not progress while on or within 8 weeks from the day of the last platinum administration.
     * Patients must have with high-grade serous or endometroid ovarian, fallopian tube, or primary peritoneal cancer. Patients must have experienced a response lasting at least 6 months to first-line platinum-based therapy but currently considered to have platinum-resistant disease per investigator's assessment (e.g, patient is not eligible for further platinum containing treatment). Patients may have had up to 4 lines of cytotoxic therapy for advanced or metastatic cancer. Neoadjuvant, adjuvant, and the combination of both will be considered as one line of therapy.
* Archival tumor tissue available or a fresh biopsy must be obtained prior to study treatment initiation
* Measurable lesions by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) 0 or 1
* Adequate organ function
* Able to take oral medications
* Female patient, if of childbearing potential, has a negative serum pregnancy test within 72 hours of taking study medication and agrees to abstain from activities that could result in pregnancy from enrollment through 120 days after the last dose of study treatment
* Male patient agrees to use an adequate method of contraception

Main Exclusion Criteria:

* Patients with primary platinum refractory ovarian cancer (ie, progressive disease on or within 6 months of first-line platinum therapy)
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis Note: Patients previously treated for brain metastases may be able to participate provided they are stable
* Patient has a known additional malignancy that progressed or required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
* Poor medical risk
* Condition (such as transfusion dependent anemia or thrombocytopenia), therapy, or laboratory abnormality that might confound the study results, or interfere with the patient's participation for the full duration of the study treatment.
* Pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study
* Immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Known active hepatitis B or hepatitis C
* Active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Prior treatment with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Prior treatment with a known poly(ADP-ribose) polymerase (PARP) inhibitor
* Heart-rate corrected QT interval (QTc) prolongation > 470 msec at screening
* Known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (28):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farkkila A, Gulhan DC, Casado J, Jacobson CA, Nguyen H, Kochupurakkal B, Maliga Z, Yapp C, Chen YA, Schapiro D, Zhou Y, Graham JR, Dezube BJ, Munster P, Santagata S, Garcia E, Rodig S, Lako A, Chowdhury D, Shapiro GI, Matulonis UA, Park PJ, Hautaniemi S, Sorger PK, Swisher EM, D'Andrea AD, Konstantinopoulos PA. Immunogenomic profiling determines responses to combined PARP and PD-1 inhibition in ovarian cancer. Nat Commun. 2020 Mar 19;11(1):1459. doi: 10.1038/s41467-020-15315-8. PMID 32193378
- [Derived] Konstantinopoulos PA, Waggoner S, Vidal GA, Mita M, Moroney JW, Holloway R, Van Le L, Sachdev JC, Chapman-Davis E, Colon-Otero G, Penson RT, Matulonis UA, Kim YB, Moore KN, Swisher EM, Farkkila A, D'Andrea A, Stringer-Reasor E, Wang J, Buerstatte N, Arora S, Graham JR, Bobilev D, Dezube BJ, Munster P. Single-Arm Phases 1 and 2 Trial of Niraparib in Combination With Pembrolizumab in Patients With Recurrent Platinum-Resistant Ovarian Carcinoma. JAMA Oncol. 2019 Aug 1;5(8):1141-1149. doi: 10.1001/jamaoncol.2019.1048. PMID 31194228
- [Derived] Vinayak S, Tolaney SM, Schwartzberg L, Mita M, McCann G, Tan AR, Wahner-Hendrickson AE, Forero A, Anders C, Wulf GM, Dillon P, Lynce F, Zarwan C, Erban JK, Zhou Y, Buerstatte N, Graham JR, Arora S, Dezube BJ, Telli ML. Open-label Clinical Trial of Niraparib Combined With Pembrolizumab for Treatment of Advanced or Metastatic Triple-Negative Breast Cancer. JAMA Oncol. 2019 Aug 1;5(8):1132-1140. doi: 10.1001/jamaoncol.2019.1029. PMID 31194225

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted in the United States.
Pre-assignment Details: A total of 122 participants (14 in Phase 1 and 108 in Phase 2) were enrolled in the study (Safety analysis set included all participants who received any amount of study treatment in Phase 1 or Phase 2).
Groups:
- Phase 1: Niraparib 200 mg + Pembrolizumab: Participants received Niraparib 200 milligrams (mg) orally once daily from Days 1 to 21 and Pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle.
- Phase 1: Niraparib 300 mg + Pembrolizumab: Participants received Niraparib 300 mg orally once daily from Days 1 to 21 and Pembrolizumab 200 mg IV on Day 1 of each 21-day cycle.
- Phase 2 OC: Niraparib 200mg + Pembrolizumab: Participants with Ovarian Cancer (OC) received recommended phase 2 dose (RP2D) of Niraparib 200 mg orally once daily and Pembrolizumab 200 mg IV on Day 1 of each 21-day cycle.
- Phase 2 TNBC: Niraparib 200mg + Pembrolizumab: Participants with Triple Negative Breast Cancer (TNBC) received RP2D of Niraparib 200 mg orally once daily and Pembrolizumab 200 mg IV on Day 1 of each 21-day cycle.
Period: Phase 1: (Up to a Maximum of 22 Months)
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab | Phase 2 OC: Niraparib 200mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Started | 7 | 7 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 0 | 0
Not completed — Death | 5 | 5 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Sponsor decision | 0 | 1 | 0 | 0
Not completed — Radiologic Disease Progression | 0 | 1 | 0 | 0
Period: Phase 2: (Up to a Maximum of 54 Months)
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab | Phase 2 OC: Niraparib 200mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Started | 0 | 0 | 53 | 55
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 53 | 55
Not completed — Death | 0 | 0 | 30 | 42
Not completed — Lost to Follow-up | 0 | 0 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 2
Not completed — Sponsor decision | 0 | 0 | 2 | 2
Not completed — Radiologic Disease Progression | 0 | 0 | 6 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Participant request | 0 | 0 | 2 | 1
Not completed — Participants went on Rollover Study | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The Baseline analysis Population consisted of all participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab | Phase 2 OC: Niraparib 200mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab | Total
Number analyzed (Participants) | 7 | 7 | 53 | 55 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 37 | 47 | 92
  >=65 years | 3 | 3 | 16 | 8 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 53 | 55 | 122
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 3 | 3 | 7
  Not Hispanic or Latino | 6 | 6 | 50 | 51 | 113
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 8 | 9
  White | 7 | 7 | 46 | 43 | 103
  More than one race | NA — Data on multiple race categories not collected | NA — Data on multiple race categories not collected | NA — Data on multiple race categories not collected | NA — Data on multiple race categories not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 0 | 0 | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 53 | 55 | 122

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Reporting Dose-Limiting Toxicities (DLTs)
Description: DLTs are defined as: Any treatment-related Grade >=3 non-hematologic clinical (non-laboratory) adverse event (AE); Any treatment-related Grade 3 or Grade 4 non-hematologic laboratory (lab) abnormality if Medical intervention is required to treat the participant or the abnormality leads to hospitalization or the abnormality persists for >=7 days; Any treatment-related hematologic toxicity specifically defined as: Thrombocytopenia Grade 4 for >=7 days, or Grade 3 or 4 associated with bleeding or requiring platelet transfusion, Neutropenia Grade 4 for >=7 days, or Grade 3 or 4 associated with infection or febrile neutropenia, Anemia Grade 4, or Grade 3 or 4 requiring blood transfusion; Any treatment-related AE leading to niraparib dose interruption per the following criteria: A dose interruption for a non-DLT lab abnormality lasting >=14 days, A dose in interruption per dose modification rules for non-hematologic AE leading to <80 percent (%) of an intended dose being administered.
Time Frame: During Cycle 1, ie, during the first 21 days of treatment
Population: DLT Analysis Set comprised of all Phase 1 participants who completed the first cycle of therapy. The assessment of DLTs in Phase 1 included only those participants completing the first cycle of therapy, unless the participant discontinued study drug due to a DLT. Only those participants with data available at specified data point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) as Measured by Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1
Description: ORR is defined as the percentage of participants with a confirmed best overall response of Complete Response (CR) or Partial Response (PR), RECIST v1.1 for target lesions as assessed by the Investigator. CR is defined as disappearance of all target lesions, Any pathological lymph nodes must be <10 millimeters (mm) in the short axis; PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: Up to 40 weeks
Population: Full Analysis Set comprised of all Phase 2 participants who received any amount of study treatment. Only those participants with data available at specified time points were analyzed. .
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 OC: Niraparib 200mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Number analyzed (Participants) | 53 | 55
Percentage of participants | 15.1 [7.7 to 25.6] | 18.2 [10.2 to 28.9]

3. Secondary Outcome: Phase 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event was any untoward medical occurrence that occurs in a participant or clinical investigation participant administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with this treatment. TEAEs were any new AE that begins, or any pre-existing condition that worsens in severity, after at least 1 dose of study treatment has been administered.
Time Frame: Up to a maximum of 22 months
Population: Safety Analysis Set comprised of all participants who received any amount of study treatment in Phase 1 or Phase 2. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 7 | 7
Participants | 7 | 7

4. Secondary Outcome: Phase 2: Number of Participants With TEAEs
Description: as for outcome 3
Time Frame: Up to a maximum of 54 months
Population: Safety Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 OC: Niraparib 200 mg + Pembrolizumab: Participants with Ovarian Cancer (OC) received recommended phase 2 dose (RP2D) of Niraparib 200 mg orally once daily and Pembrolizumab 200 mg IV on Day 1 of each 21-day cycle.
- Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab: Participants with Triple Negative Breast Cancer (TNBC) received RP2D of Niraparib 200 mg orally once daily and Pembrolizumab 200 mg IV on Day 1 of each 21-day cycle.
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab
Number analyzed (Participants) | 53 | 55
Participants | 53 | 54

5. Secondary Outcome: Phase 2: Overall Response Rate (ORR) as Measured by Immune-related RECIST (irRECIST)
Description: ORR by irRECIST is defined as the percentage of participants with a confirmed best overall response of CR or PR using irRECIST. Immune related complete response (irCR) is defined as at least two radiographic determinations of CR, at least 4 weeks apart and before Immune related progressive disease (irPD - defined as at least two consecutive radiographic determinations of progressive disease [PD] at least 4 weeks apart) at least 4 weeks apart. Immune related partial response (irPR) defined as at least two radiographic determinations of PR or better at least 4 weeks apart and before irPD (and not qualifying for an irCR).
Time Frame: Up to a maximum of 54 months
Population: Full Analysis Set. IrRECIST data were invalid due to errors in the collection approach. Hence, data for this outcome measure were not reported. This decision was documented in the final Statistical Analysis Plan (SAP) (Version 2, 21-March-2019) and approved before database lock which occurred on 22-October-2021.
Arm/Group | Phase 2 OC: Niraparib 200mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase 2: Duration of Response (DOR) as Measured by RECIST v1.1
Description: DoR per RECIST v1.1 was defined as the time from first documented evidence of CR or PR until first documented disease progression per RECIST v1.1 based upon investigator assessment or death due to any cause, whichever occurs first, among participants who demonstrated CR or PR as the best overall response per RECIST v1.1. CR is defined as disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeters (mm) in the short axis. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: Up to a maximum of 54 months
Population: Full Analysis Set. Only those participants with data available at specified time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab
Number analyzed (Participants) | 8 | 10
Months | 14.4 [8.3 to 18.7] | 21.5 [8.4 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived.

7. Secondary Outcome: Phase 2: DOR as Measured by irRECIST
Description: DOR was defined as the time from the initial response (irCR, irPR or irSD) to progression or death, whichever occurs first. Response was to be assessed using the irRECIST. Immune related complete response (irCR) is at least two radiographic determinations of CR at least 4 weeks apart and before Immune related progressive disease (irPD - defined as at least two consecutive radiographic determinations of PD at least 4 weeks apart) at least 4 weeks apart. Immune related partial response (irPR) defined as at least two radiographic determinations of PR or better at least 4 weeks apart and before irPD (and not qualifying for an irCR).
Time Frame: Up to a maximum of 54 months
Population: as for outcome 5
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Phase 2: Disease Control Rate (DCR) as Measured by RECIST v1.1
Description: DCR is defined as the percentage of participants who achieved a CR or PR or stable disease (SD) using RECIST (v1.1) as assessed by the investigator.
Time Frame: Up to 40 weeks
Population: Full Analysis Set. Only those participants with data available at specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2 OC: Niraparib 200mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Number analyzed (Participants) | 53 | 55
Percentage of participants | 58.5 [46.3 to 70.0] | 41.8 [30.5 to 53.8]

9. Secondary Outcome: Phase 2: DCR as Measured by irRECIST
Description: DCR is percentage of participants achieving best overall response of confirmed irCR, irPR, or immune-related stable disease (irSD) (lasting at least 5 weeks), according to irRECIST from the first dose date until disease progression/recurrence.
Time Frame: Up to a maximum of 54 months
Population: as for outcome 5
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 2: Progression Free Survival (PFS) as Measured by RECIST v1.1
Description: PFS is defined as the time from first dose of study treatment to the earlier date of assessment of progression or death by any cause in the absence of progression based on the time of first documentation of disease progression per RECIST v1.1. Progression is defined using RECIST v1.1 as a 20% increase in the sum of the diameter of target lesions or unequivocal progression of existing non-target lesions or the appearance of one or more new lesions.
Time Frame: Up to a maximum of 54 months
Population: Full Analysis Set. Only those participants with data available at specified time point were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab
Number analyzed (Participants) | 53 | 55
Months | 3.4 [2.1 to 8.2] | 2.5 [1.4 to 6.4]

11. Secondary Outcome: Phase 2: PFS as Measured by irRECIST
Description: Progression free survival is defined as the duration of time from the date of study enrollment until time of disease relapse, disease progression, or death, whichever comes first. Progression was to be assessed using the Immune Related Response Evaluation Criteria in Solid Tumors (irRECIST). Immune related progressive disease (irPD) is defined as at least two consecutive radiographic determinations of progressive disease (PD - e.g., appearance of one or more new lesions) at least 4 weeks apart).
Time Frame: Up to a maximum of 54 months
Population: as for outcome 5
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the time from date of first dose of study treatment to the date of death by any cause.
Time Frame: Up to a maximum of 54 months
Population: Full Analysis Set. Only those participants with data available at specified time point were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Number analyzed (Participants) | 53 | 55
Months | 17.1 [7.9 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third-quartile could not be derived. | 9.4 [3.2 to 22.2]

13. Secondary Outcome: Phase 1: Area Under the Plasma Concentration-time Curve From Time 0 (Predose) to 24 Hours Post Dose (AUC [0-24]) of Niraparib
Description: Blood samples were collected at indicated time points. Pharmacokinetic (PK) analysis of Niraparib was conducted using standard non-compartmental analysis.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set comprised of all participants with sufficient data to enable estimation of at least one PK parameter. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour*nanogram per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 6 | 6
Hour*nanogram per milliliter | 6524.035 (2606.263) | 8855.687 (1415.318)

14. Secondary Outcome: Phase 1: AUC (0-24) of Major Metabolite of Niraparib (M1)
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of major metabolite of Niraparib (M1) was conducted using standard non-compartmental analysis.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour*nanogram per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 3 | 2
Hour*nanogram per milliliter | 4886.115 (975.011) | 11076.538 (6691.358)

15. Secondary Outcome: Phase 1: Minimum Observed Plasma Concentration (Cmin) and Maximum Observed Plasma Concentration (Cmax) of Niraparib
Description: Blood samples were collected at indicated time points. Pharmacokinetic analysis of Niraparib was conducted using standard non-compartmental analysis.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 7 | 7
Nanogram per milliliter
  Cmin | 174.00 (84.922) | 205.63 (196.714)
  Cmax | 546.0 (195.95) | 711.3 (189.98)

16. Secondary Outcome: Phase 1: Cmin and Cmax of Major Metabolite of Niraparib (M1)
Description: as for outcome 14
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 7 | 7
Nanogram per milliliter
  Cmin | 42.114 (42.765) | 46.677 (45.343)
  Cmax | 340.14 (89.356) | 491.66 (226.122)

17. Secondary Outcome: Phase 1: Apparent Oral Clearance (CL/F) of Niraparib
Description: Blood samples were planned to be collected for to determine CL/F of Niraparib.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. The current PK sampling schedule made the estimation of CL/F incalculable due to long half life of Niraparib.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 7 | 7
Liters per hour | NA (NA) — NA indicates that data was not available as the current PK sampling schedule made the estimation of CL/F incalculable due to long half-life of Niraparib. | NA (NA) — NA indicates that data was not available as the current PK sampling schedule made the estimation of CL/F incalculable due to long half-life of Niraparib.

18. Secondary Outcome: Phase 1: Apparent Oral Clearance (CL/F) of Major Metabolite of Niraparib (M1)
Description: Blood samples were planned to be collected for to determine CL/F of major metabolite (M1) of Niraparib.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. The current PK sampling schedule made the estimation of CL/F incalculable due to long half life of major metabolite of Niraparib (M1).
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 7 | 7
Liters per hour | NA (NA) — NA indicates that data was not available as the current PK sampling schedule made the estimation of CL/F incalculable due to long half-life of major metabolite of Niraparib (M1). | NA (NA) — NA indicates that data was not available as the current PK sampling schedule made the estimation of CL/F incalculable due to long half-life of major metabolite of Niraparib (M1).

19. Secondary Outcome: Phase 1: Volume of Distribution (Vz/F) of Niraparib
Description: Blood samples were planned to be collected for to determine Vz/F of Niraparib.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. The current PK sampling schedule made the estimation of Vz/F incalculable due to long half life of Niraparib.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 7 | 7
Liters | NA (NA) — NA indicates that data was not available the current PK sampling schedule made the estimation of Vz/F incalculable due to long half-life of Niraparib. | NA (NA) — NA indicates that data was not available the current PK sampling schedule made the estimation of Vz/F incalculable due to long half-life of Niraparib.

20. Secondary Outcome: Phase 1: Volume of Distribution (Vz/F) of Major Metabolite of Niraparib (M1)
Description: Blood samples were planned to be collected for to determine Vz/F of major metabolite (M1) of Niraparib.
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 1 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. The current PK sampling schedule made the estimation of Vz/F incalculable due to long half life of major metabolite of Niraparib (M1).
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 7 | 7
Liters | NA (NA) — NA indicates that data was not available as the current PK sampling schedule made the estimation of Vz/F incalculable due to long half-life of major metabolite of Niraparib (M1). | NA (NA) — NA indicates that data was not available as the current PK sampling schedule made the estimation of Vz/F incalculable due to long half-life of major metabolite of Niraparib (M1).

21. Secondary Outcome: Phase 1: AUC at Steady State (AUC,ss) of Niraparib
Description: as for outcome 15
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 2 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour*nanograms per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 4 | 2
Hour*nanograms per milliliter | 27396.910 (15097.186) | 30799.742 (9868.734)

22. Secondary Outcome: Phase 1: AUC,ss of Major Metabolite of Niraparib (M1)
Description: as for outcome 14
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 2 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hour*nanograms per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 1 | 1
Hour*nanograms per milliliter | 32878.205 (NA) — NA indicates that standard deviation could not be calculated for single participant. | 127430.14 (NA) — NA indicates that standard deviation could not be calculated for single participant.

23. Secondary Outcome: Phase 1: Minimum Observed Plasma Concentration at Steady State (Cmin,ss) and Maximum Observed Plasma Concentration at Steady State (Cmax,ss) of Niraparib
Description: as for outcome 15
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 2 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 4 | 3
Nanograms per milliliter
  Cmin,ss | 878.75 (651.122) | 849.00 (194.841)
  Cmax,ss | 1585.5 (812.63) | 1606.7 (261.02)

24. Secondary Outcome: Phase 1: Cmin,ss and Cmax,ss of Major Metabolite of Niraparib (M1)
Description: as for outcome 14
Time Frame: Pre-dose and 1, 2, 4, 6, 8, 24 Hours post-dose on Cycle 2 Day 1(each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab
Number analyzed (Participants) | 4 | 3
Nanograms per milliliter
  Cmin,ss | 1410.000 (207.686) | 3280.000 (1460.411)
  Cmax,ss | 2177.50 (475.000) | 4213.33 (1515.333)

25. Secondary Outcome: Phase 2: Plasma Concentrations of Niraparib
Description: Blood samples were collected by sparse PK sampling to analyze plasma concentration of Niraparib.
Time Frame: Pre-dose and 2 Hours post-dose on Cycle 1 Day 1; Pre-dose and 2 Hours post-dose on Cycle 2 Day 1(each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Number analyzed (Participants) | 50 | 54
Nanograms per milliliter
  Cycle 1 Day 1: Predose: number analyzed (Participants) | 49 | 51
  Cycle 1 Day 1: Predose | 0.000 (0.000) | 0.000 (0.000)
  Cycle 1 Day 1; 2 hours post dose: number analyzed (Participants) | 48 | 52
  Cycle 1 Day 1; 2 hours post dose | 315.979 (199.798) | 302.642 (267.128)
  Cycle 2 Day 1; Predose: number analyzed (Participants) | 27 | 26
  Cycle 2 Day 1; Predose | 441.978 (229.948) | 510.154 (263.634)
  Cycle 2; Day 1; 2 hours post dose: number analyzed (Participants) | 28 | 27
  Cycle 2; Day 1; 2 hours post dose | 764.500 (370.140) | 884.185 (508.607)

26. Secondary Outcome: Phase 2: Plasma Concentrations of Major Metabolite of Niraparib (M1)
Description: Blood samples were collected by sparse PK sampling to analyze plasma concentration of major metabolite of Niraparib (M1).
Time Frame: Pre-dose and 2 Hours post-dose on Cycle 1 Day 1; Pre-dose and 2 Hours post-dose on Cycle 2 Day 1 (each cycle of 21 days)
Population: Pharmacokinetic Analysis Set. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200mg + Pembrolizumab
Number analyzed (Participants) | 50 | 54
Nanograms per milliliter
  Cycle 1 Day 1; Predose: number analyzed (Participants) | 49 | 51
  Cycle 1 Day 1; Predose | 0.000 (0.000) | 0.000 (0.000)
  Cycle 1 Day1; 2 hours post dose: number analyzed (Participants) | 48 | 52
  Cycle 1 Day1; 2 hours post dose | 116.666 (89.108) | 84.875 (92.206)
  Cycle 2 Day 1; Predose: number analyzed (Participants) | 27 | 26
  Cycle 2 Day 1; Predose | 1278.926 (625.932) | 1070.923 (648.225)
  Cycle 2 Day 1; 2 hours post dose: number analyzed (Participants) | 28 | 27
  Cycle 2 Day 1; 2 hours post dose | 1500.143 (976.572) | 1205.444 (858.698)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAE) and non-serious adverse events (non-SAEs) were collected up to a maximum of 22 months in Phase 1 and up to a maximum of 54 months in Phase 2 of the study
Description: All-cause mortality, SAE and non-SAE were collected in Safety analysis set which comprised of all participants who received any amount of study treatment in Phase 1 or Phase 2.
Arm/Group | Phase 1: Niraparib 200 mg + Pembrolizumab | Phase 1: Niraparib 300 mg + Pembrolizumab | Phase 2 OC: Niraparib 200 mg + Pembrolizumab | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/7 | 5/7 | 30/53 | 42/55
Serious Adverse Events (participants affected / at risk) | 6/7 | 4/7 | 22/53 | 24/55
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 52/53 | 54/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Niraparib 200 mg + Pembrolizumab (N=7) | Phase 1: Niraparib 300 mg + Pembrolizumab (N=7) | Phase 2 OC: Niraparib 200 mg + Pembrolizumab (N=53) | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab (N=55)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 4
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 5 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 4 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 3
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 3
Stoma site infection (Infections and infestations) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 3
Mental status changes (Psychiatric disorders) | 1 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Niraparib 200 mg + Pembrolizumab (N=7) | Phase 1: Niraparib 300 mg + Pembrolizumab (N=7) | Phase 2 OC: Niraparib 200 mg + Pembrolizumab (N=53) | Phase 2 TNBC: Niraparib 200 mg + Pembrolizumab (N=55)
Anaemia (Blood and lymphatic system disorders) | 5 | 5 | 19 | 24
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 14 | 14
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 3
Hypothyroidism (Endocrine disorders) | 2 | 0 | 7 | 8
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 13 | 8
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 5 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 2 | 28 | 24
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 15 | 13
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 4 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 5 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 32 | 34
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 3 | 4
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 21 | 13
Asthenia (General disorders) | 0 | 0 | 3 | 0
Chills (General disorders) | 0 | 0 | 3 | 0
Fatigue (General disorders) | 4 | 3 | 32 | 30
Swelling (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 3 | 1 | 0 | 6
Pain (General disorders) | 0 | 0 | 0 | 4
Peripheral swelling (General disorders) | 0 | 1 | 4 | 0
Pyrexia (General disorders) | 0 | 0 | 7 | 4
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 5
Sinusitis (Infections and infestations) | 0 | 0 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 6
Urinary tract infection (Infections and infestations) | 0 | 0 | 7 | 10
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 3
Alanine aminotransferase increased (Investigations) | 0 | 0 | 8 | 11
Amylase increased (Investigations) | 0 | 0 | 4 | 0
Anticoagulation drug level increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 8 | 15
Blood alkaline phosphatase decreased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 6 | 9
Blood creatinine increased (Investigations) | 0 | 0 | 4 | 4
Creatinine renal clearance increased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 3
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 10
Neutrophil count decreased (Investigations) | 0 | 0 | 7 | 6
Platelet count decreased (Investigations) | 0 | 2 | 7 | 9
Troponin increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 8 | 3
White blood cell count decreased (Investigations) | 1 | 1 | 4 | 8
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 17 | 15
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 6 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 5 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 7 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 1 | 7 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 8 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 8 | 11
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 7
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 7 | 6
Dysgeusia (Nervous system disorders) | 1 | 3 | 4 | 5
Headache (Nervous system disorders) | 2 | 2 | 14 | 14
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 3 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 3 | 8
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 11 | 14
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 9 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 11 | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 8 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 7 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 7
Hypertension (Vascular disorders) | 0 | 0 | 5 | 5
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 4
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Flushing (Vascular disorders) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT02657889/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT02657889/SAP_001.pdf